CLINICAL TRIAL: NCT04680026
Title: A Phase 2, Two-Stage, Serial Cohort Dose Escalation and Expansion Study of a Single Intravenous Infusion of HBI 3000 for the Conversion of Atrial Fibrillation (AF) of Recent Onset
Brief Title: A Study of IV HBI-3000 for the Conversion Recent Onset Atrial Fibrillation (AF)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: HUYABIO International, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HBI-3000-402
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation
Keywords: cardioversion
MeSH Terms: conditions — Atrial Fibrillation | interventions — sulcardine sulfate

STUDY DESIGN:
Intervention Model Description: Allocation: Stage A: non-randomized; Stage B: randomized, double-blind and placebo-controlled Intervention Model: Two-stage study Masking: None; Stage A (open label); Stage B: randomized, double-blind and placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Drug: HBI-3000, Stage A Dose Level 1 (Experimental): Stage A Open Label HBI-3000 Dose Level 1: 200 mg
  Interventions: Drug: HBI-3000
- Drug: HBI-3000, Stage A Dose Level 2 (Experimental): Stage A Open Label HBI-3000 Dose Level 2: 350 mg planned
  Interventions: Drug: HBI-3000
- Drug: HBI-3000, Stage A Dose Level 3 (Experimental): Stage A Open Label HBI-3000 Dose Level 2: 500 mg planned
  Interventions: Drug: HBI-3000
- Drug: HBI-3000, Stage B Dose Level 1 (Experimental): Stage B Double-blind placebo controlled, Cohort 1 HBI-3000 Dose Level 1: Selected based on Stage A results
  Interventions: Drug: HBI-3000; Drug: Placebo
- Drug: HBI-3000, Stage B Dose Level 2 (Experimental): Stage B Double-blind placebo controlled, Cohort 2 HBI-3000 Dose Level 2: Selected based on Stage A, and Stage B Cohort 1 results
  Interventions: Drug: HBI-3000; Drug: Placebo

INTERVENTIONS:
Drug: HBI-3000 — Small molecule, multi-ion channel blocker
  Other Names: sulcardine sulfate
Drug: Placebo — Normal saline
  Arms: Drug: HBI-3000, Stage B Dose Level 1; Drug: HBI-3000, Stage B Dose Level 2

SUMMARY:
This Phase 2 study is a two-stage, serial cohort dose escalation and expansion study of a single 30-minute (IV) infusion of HBI-3000 for the conversion of patients with recent-onset atrial fibrillation (AF).

Stage A is open label and all patients will receive HBI-3000. In each of three dose cohorts, up to 10 patients will receive HBI-3000 by IV infusion (30 minutes). Three different dose levels are planned to be administered serially, lowest to highest, with assessment of safety, tolerability, and efficacy prior to proceeding to the next dose level group.

Following Stage A, the iDMC will recommend up to two doses of HBI-3000 to be further explored in Stage B. Stage B is a serial, randomized, double-blind and placebo-controlled cohort of two different doses of HBI-3000, with a dose decision after the first cohort. Stage B will be powered to show a difference between HBI-3000 and placebo in conversion rate at each of the two dose levels.

DETAILED DESCRIPTION:
This is a two-stage study in patients with AF of recent onset:

Stage A is open label and all patients will receive HBI-3000. In each of three dose cohorts, up to 10 patients will receive HBI-3000 by IV infusion (30 minutes). For each dosing cohort, sentinel dosing is planned. Each patient may enroll only once in the study, will be enrolled into only one dose cohort and receive only a single dose treatment. In Stage A, three different dose levels are planned to be administered serially, lowest to highest, with assessment of safety, tolerability, and efficacy prior to proceeding to the next dose level group. The actual dose levels may be modified, and additional dose levels may be considered based on the observed results at each cohort.

Stage B is the randomized, double-blind and placebo-controlled part of the study. Study drug for Stage B patients is either HBI-3000 or placebo. Two cohorts will be enrolled sequentially, lowest dose level first, with safety, efficacy, and available PK results evaluated by the Sponsor and iDMC prior to enrolling patients in the next/higher dose cohort. The dose level for the second cohort may be adjusted following interim review of results in the first cohort. Patients will be randomized to receive a single IV infusion of HBI 3000 or placebo over 30 minutes. In each of the dose cohorts, sequentially enrolled patients will be randomized at 2:1 ratio so that 40 patients will receive HBI 3000 infusion and 20 patients will receive placebo infusion. Each patient may enroll only once in the study, will be enrolled into only one dose cohort and receive only a single dose treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years of age
* Sustained AF of > 2 hours and < 72 hours duration
* Eligible for cardioversion (electrical and pharmacologic)
* On adequate anticoagulant therapy or eligible for anticoagulation during treatment and for at least 30 days duration after treatment if indicated by ACC/AHA/HRS or country specific national or international guidelines for thromboembolic risk reduction related to AF

Exclusion Criteria:

* Atrial fibrillation < 2 hours or > 72 hours duration or with duration not reliably established at the time of dosing
* Hemodynamic instability that may require emergency electrical cardioversion
* Atrial flutter
* Moderate to severe HF
* Clinical or ECG signs of acute cardiac ischemia or digitalis toxicity
* Known or suspected hyperthyroidism
* Cardiac surgery, stroke, TIA, acute MI/ PCI, unstable angina, or persistent angina at rest within the previous 3 months
* Presence of LA thrombus by TEE or TTE
* Presence of concurrent myocarditis or endocarditis
* ECG abnormalities: Current QTcF > 480 msec; QRS interval > 120 msec and/or a complete bundle branch block (BBB)l Delta wave or other pre-excitation pattern consistent with WPW syndrome; Acute coronary ischemia patterns
* Use of medication that prolongs the QTc interval or history of: Long QT syndrome, congenital or acquired; Torsades de Pointes (TdP); Brugada Syndrome; Ventricular arrhythmia (not including infrequent isolated PVC)
* Concurrent treatment with Class I or III antiarrhythmic drugs, metformin or strong CYP2D6 inhibitors (unless the medication is discontinued > 5 half-lives before enrollment)
* Treatment with oral amiodarone in the previous 3 months or IV amiodarone administered within 24 hours prior to planned Study Drug administration
* Use of vernakalant, or any experimental drug within 30 days or five half-lives (whichever is longer) of Study Drug administration, or use of an invasive investigational medical device within 2 months prior to Study Drug administration, or current enrollment in another study with investigational agent or procedure
* Clinically significant laboratory abnormalities

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of intravenously (IV) administered HBI-3000 in patients with Atrial Fibrillation (AF) of recent onset, as measured by the incidence of adverse events (AEs) | 30 days
  Evaluate the safety of intravenously (IV) administered HBI-3000 in patients with Atrial Fibrillation (AF) of recent onset, as measured by the incidence of adverse events (AEs)
Evaluate the safety of intravenously (IV) administered HBI-3000 in patients with Atrial Fibrillation (AF) of recent onset, as measured by changes in heart rate (HR) | 90 minutes
  Evaluate the safety of intravenously (IV) administered HBI-3000 in patients with Atrial Fibrillation (AF) of recent onset, as measured by change in heart rate (HR) from baseline (prior to Study Drug infusion) to study timepoints during and after Study Drug infusion, specifically:
  HR < 40 bpm for 2 minutes or longer within 90 minutes of initiation of the infusion
  HR increase > 25 percent before conversion to SR (based on one minute averages compared between the event and the first minute of stable telemetry)
  HR > 120 bpm for one minute or longer after conversion to SR and within 90 minutes of initiation of the infusion
Evaluate the safety of intravenously (IV) administered HBI-3000 in patients with Atrial Fibrillation (AF) of recent onset, as measured by change in blood pressure (BP) | 90 minutes
  Evaluate the safety of intravenously (IV) administered HBI-3000 in patients with Atrial Fibrillation (AF) of recent onset, as measured by changes in blood pressure (BP) from baseline (prior to Study Drug infusion) to study timepoints during and after Study Drug infusion, specifically: Systolic BP < 90 mmHg for > 1 minute during SR and within 90 minutes of initiation of the infusion
Evaluate the safety of intravenously (IV) administered HBI-3000 in patients with Atrial Fibrillation (AF) of recent onset, as measured by ECG interval changes above a specific level | 24 hours
  Evaluate the safety of intravenously (IV) administered HBI-3000 in patients with Atrial Fibrillation (AF) of recent onset, as measured by ECG interval changes from baseline (prior to Study Drug infusion) to 24 hour post-infusion, specifically:
  QTcF: > 500 msec and > 60 msec above the 24-hour post-conversion level during SR
  PR: > 50 percent above the 24-hour post-conversion level during SR
  QRS: ≥ 33 percent above the 24-hour post-conversion level during SR
The efficacy of intravenously (IV) administered HBI-3000 as measured by the proportion of patients with AF of recent onset who convert to SR | 120 minutes
  Evaluate the efficacy of intravenously (IV) administered HBI-3000 in patients with Atrial Fibrillation (AF) of recent onset as measured by the proportion of patients with AF of recent onset who convert to SR (for a duration of at least one minute) within 120 minutes of the start of infusion

SECONDARY OUTCOMES:
Evaluate the time to conversion to SR from start of infusion | 24 hours
  Efficacy as measured by the time from the start of infusion to the time of conversion to SR for a duration of at least one minute
Evaluate the proportion of patients with sustained AF or late conversion to SR | 12 hours, 24 hours and 7 days
  Efficacy as measured by the proportion of patients with sustained or late conversion of AF of recent onset to SR at 12 hours, 24 hours and 7 days after start of infusion

CONTACTS AND LOCATIONS:
Locations (14):
- United States (4):
  - NCH Research Institute, Naples, Florida
  - Prairie Education & Research, Springfield, Illinois
  - North Mississippi Medical Center, Tupelo, Mississippi
  - CHRISTUS Trinity Mother Frances Hospital - Tyler, Tyler, Texas
- University Clinical Center of the Republic of Srpska, Banja Luka, Bosnia and Herzegovina
- Canada (3):
  - Montreal Heart Institute, Montreal, Quebec
  - Centre hospitalier de L'Universite de Montral (CHUM), Montreal, Quebec
  - Centre integre de sante et de services sociaux de Lanaudiere - Hopital Pierre-Le Gardeur, Terrebonne, Quebec
- New Zealand (2):
  - Waikato Hospital, Hamilton
  - Wellington Regional Hospital, Wellington
- Serbia (4):
  - Niš University Clinical Center, Niš, Bulevar Doktora
  - University Clinical Center of Serbia, Belgrade
  - Dedinje Institute for Cardiovascular Diseases, Belgrade
  - University Hospital Medical Center Bezanijska kosa, Belgrade

IPD SHARING:
Plan to Share IPD: No